CLINICAL TRIAL: NCT03222206
Title: The Comparison of Effect Between Salsalate and Placebo in Osteoarthritis With Nonalcoholic Fatty Liver Disease: Investigator Initiated Randomized Placebo-controlled Double-blind, Pilot Study
Brief Title: The Comparison of Effect Between Salsalate and Placebo in Osteoarthritis With Nonalcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Kuhnil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Ji Hoon Kim, Associate professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KUGH16353
Record Dates: First submitted 2017-07-08; First posted 2017-07-19 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Non Alcoholic Fatty Liver; Osteo Arthritis
Keywords: Hepatokine; Adipokine; Saccharometabolism; Lipid metabolism
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — salicylsalicylic acid

STUDY DESIGN:
Intervention Model Description: Salsalate (2g/d), Place (2g/d)
Who Masked: Participant, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salsalate (Experimental): 17 patients received continuous medication with salsalate 2g/day after run-in period
  Interventions: Drug: Salsalate
- Placebo (Placebo Comparator): 17 patients received continuous medication with Placebo 2g/day after run-in period
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Salsalate — 1. Medicate salsalate 2g/day after run-in period
  2. Check side effect after 1 month and Control dosage (2g/day or 3g/day)
  3. Check side effect after 2 month
  Other Names: A03850041
  Arms: Salsalate
Other: Placebo — 1. Medicate placebo 2g/day after run-in period
  2. Check side effect after 1 month and Control dosage (2g/day or 3g/day)
  3. Check side effect after 2 month
  Arms: Placebo

SUMMARY:
This Study purpose to verify change of variety factors that the cause of nonalcoholic fatty liver disease and its process through salsalate injection to osteoarthritis patient who has non alcoholic fatty liver

DETAILED DESCRIPTION:
Salsalate, the salicylic acid dimer that is one of anti-inflammatory and kind of salicylate. Aspirin(Acetylated salicylic) is known as nonsteroidal anti-inflammatory, also salsalate is widely used painkiller and anti-inflammatory without prescription in Europe and America through the long time and it was approved as osteoarthritis and rheumarthritis treatment in Korea. Especially salsalate is switched to salicylic acid(active metabolite) 15% rate lower than the same dose of aspirin (3.5g vs. 5g).

Salsalate is cyclooxygenase antagonist, it make anti-inflammatory effect by hinder creation of variety inflammatory induction factors like interleukin-6, Tumor Necrosis Factor (TNF)-alpha, C-reactive protein. This anti-inflammatory reaction is known to block Nuclear Factor(NF)-kappaB gene action by hinder action of IkappaB kinase. Also salsalate was reported it has positive effect to gluco metabolism as performed role of insulin-sensitizing. Therefore, the above mechanism of salsalate was expected that it can be had positive effect to metabolic disease like diabetes and obesity, and related studies are performed considerably at present.

There is no clinical trial for non alcoholic fatty acid related salsalate, and there was the animal study result that salsalate may reduce occurence of non alcoholic fatty acid and fibrosis by hinder non alcoholic fatty acid creation and inflammation mediation path.

Therefore, this Study purpose to verify change of variety factors that the cause of nonalcoholic fatty liver disease and its process through salsalate injection to osteoarthritis patient who has non alcoholic fatty liver

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis patient who has non alcoholic fatty liver
* Standard of non alcoholic fatty liver diagnosis

  1. Fatty liver on abdominal ultrasonography
  2. Patient who has no evidence as hepatitis B, hepatitis C, immune hepatitis, metabolic hepatitis and other chronic hepatitis
* Osteoarthritis patient who has never been treated

Exclusion Criteria:

* Unsuitable on inclusion criteria
* Thiazolidinedione injected patient for diabetes treatment or patient who has changed injected drug last 6 month
* Patient who is treating nonsteroidal antiinflammatory drugs for osteoarthritis
* Renal dysfunction : serum creatinine level 1.5mg/dl or creatinine clearance < 60ml/min
* Anamnesis of gastrointestinal tract bleeding
* Upper 5 times(200IU/l) the normality of Aspartate Transaminase(AST), Alanine Transaminase(ALT)
* Pregnant or Breastfeeding
* Patient who has untreated malignant tumor
* Liver transplantation patient
* Patient who has liver function Child-Pugh B over
* Patient who has serious disease that was estimated influence to study (e.g. Congestive heart failure, Kidney failure, Chronic pancreatitis, Malignant tumor)
* Patients who has been injected immunomodulatory and immunosuppressant(inclusive universal corticosteroids) before 6 month enrollment or at present
* Patient who was judged unsuitable for study by investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
Change of controlled attenuation parameter | baseline and 8weeks
  Estimation of salsalate single injection group and placebo injection group
Change of hepatokine as Fetuin-A | baseline and 8weeks
  Estimation of salsalate single injection group and placebo injection group
Change of pulse wave velocity | baseline and 8weeks
  Estimation of salsalate single injection group and placebo injection group
Change of adipokine as Adiponectin | baseline and 8weeks
  Estimation of salsalate single injection group and placebo injection group

SECONDARY OUTCOMES:
Change of controlled attenuation parameter | baseline and 4weeks
  Estimation of salsalate single injection group and placebo injection group
Change of hepatokine as Fetuin-A | baseline and 4weeks
  Estimation of salsalate single injection group and placebo injection group
Change of pulse wave velocity | baseline and 4weeks
  Estimation of salsalate single injection group and placebo injection group
Change of adipokine as Adiponectin | baseline and 4weeks
  Estimation of salsalate single injection group and placebo injection group
Numerical value change of fatty liver index | baseline, 4weeks and 8weeks
  Estimation of salsalate single injection group and placebo injection group
Numerical value change of hepatic fibrosis as Nonalcoholic Fatty Liver Disease(NAFLD) fibrosis score | baseline, 4weeks and 8weeks
  Estimation of salsalate single injection group and placebo injection group
Change of saccharometabolic factors as Homeostasis Model Assessment(HOMA)-Insulin Resistance(IR), Homeostasis Model Assessment(HOMA)-B, Fasting glucose, Insulin, C-peptide, HbA1c, Glycated albumin | baseline, 4weeks and 8weeks
  Estimation of salsalate single injection group and placebo injection group
Change of lipid metabolic factors as Cholesterol, Triglyceride, LDL-cholesterol HDL-cholesterol and liver function test as Aspartate Transaminase(AST) and Alanine Transaminase(ALT) | baseline, 4weeks and 8weeks
  Estimation of salsalate single injection group and placebo injection group
Change of inflammatory factors as C Reactive Protein(CRP), Tumor Necrosis Factor(TNF)-a | baseline, 4weeks and 8weeks
  Estimation of salsalate single injection group and placebo injection group
Change of liver fibrosis factors as hyaluronic acid | baseline, 4weeks and 8weeks
  Estimation of salsalate single injection group and placebo injection group
Change of symptom of osteoarthritis as visual analog score for pain | baseline, 4weeks and 8weeks
  Estimation of salsalate single injection group and placebo injection group
Change of function of osteoarthritis as WOMAC (The Western Ontario and McMaster Universities Osteoarthritis Index) | baseline, 4weeks and 8weeks
  Estimation of salsalate single injection group and placebo injection group
Stability comparison like side effect | Up to 2month
  Estimation with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Ji Hoon Kim, MD, Principal Investigator — Associate Professor
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bae JC, Cho YK, Lee WY, Seo HI, Rhee EJ, Park SE, Park CY, Oh KW, Sung KC, Kim BI. Impact of nonalcoholic fatty liver disease on insulin resistance in relation to HbA1c levels in nondiabetic subjects. Am J Gastroenterol. 2010 Nov;105(11):2389-95. doi: 10.1038/ajg.2010.275. Epub 2010 Jul 13. PMID 20628364
- [Background] Choi SY, Kim D, Kim HJ, Kang JH, Chung SJ, Park MJ, Kim YS, Kim CH, Choi SH, Kim W, Kim YJ, Yoon JH, Lee HS, Cho SH, Sung MW, Oh BH. The relation between non-alcoholic fatty liver disease and the risk of coronary heart disease in Koreans. Am J Gastroenterol. 2009 Aug;104(8):1953-60. doi: 10.1038/ajg.2009.238. Epub 2009 Jun 2. PMID 19491838
- [Background] Clark JM. The epidemiology of nonalcoholic fatty liver disease in adults. J Clin Gastroenterol. 2006 Mar;40 Suppl 1:S5-10. doi: 10.1097/01.mcg.0000168638.84840.ff. PMID 16540768
- [Background] Musso G, Cassader M, Gambino R. Diagnostic accuracy of adipose insulin resistance index and visceral adiposity index for progressive liver histology and cardiovascular risk in nonalcoholic fatty liver disease. Hepatology. 2012 Aug;56(2):788-9. doi: 10.1002/hep.25677. No abstract available. PMID 22371327
- [Background] Kim D, Choi SY, Park EH, Lee W, Kang JH, Kim W, Kim YJ, Yoon JH, Jeong SH, Lee DH, Lee HS, Larson J, Therneau TM, Kim WR. Nonalcoholic fatty liver disease is associated with coronary artery calcification. Hepatology. 2012 Aug;56(2):605-13. doi: 10.1002/hep.25593. Epub 2012 Jul 2. PMID 22271511
- [Background] Mahady SE, Webster AC, Walker S, Sanyal A, George J. The role of thiazolidinediones in non-alcoholic steatohepatitis - a systematic review and meta analysis. J Hepatol. 2011 Dec;55(6):1383-90. doi: 10.1016/j.jhep.2011.03.016. Epub 2011 Apr 14. PMID 21703200
- [Background] Aithal GP, Thomas JA, Kaye PV, Lawson A, Ryder SD, Spendlove I, Austin AS, Freeman JG, Morgan L, Webber J. Randomized, placebo-controlled trial of pioglitazone in nondiabetic subjects with nonalcoholic steatohepatitis. Gastroenterology. 2008 Oct;135(4):1176-84. doi: 10.1053/j.gastro.2008.06.047. Epub 2008 Jun 25. PMID 18718471
- [Background] Belfort R, Harrison SA, Brown K, Darland C, Finch J, Hardies J, Balas B, Gastaldelli A, Tio F, Pulcini J, Berria R, Ma JZ, Dwivedi S, Havranek R, Fincke C, DeFronzo R, Bannayan GA, Schenker S, Cusi K. A placebo-controlled trial of pioglitazone in subjects with nonalcoholic steatohepatitis. N Engl J Med. 2006 Nov 30;355(22):2297-307. doi: 10.1056/NEJMoa060326. PMID 17135584
- [Background] Klein EA, Thompson IM Jr, Tangen CM, Crowley JJ, Lucia MS, Goodman PJ, Minasian LM, Ford LG, Parnes HL, Gaziano JM, Karp DD, Lieber MM, Walther PJ, Klotz L, Parsons JK, Chin JL, Darke AK, Lippman SM, Goodman GE, Meyskens FL Jr, Baker LH. Vitamin E and the risk of prostate cancer: the Selenium and Vitamin E Cancer Prevention Trial (SELECT). JAMA. 2011 Oct 12;306(14):1549-56. doi: 10.1001/jama.2011.1437. PMID 21990298
- [Background] Kahn SE, Zinman B, Lachin JM, Haffner SM, Herman WH, Holman RR, Kravitz BG, Yu D, Heise MA, Aftring RP, Viberti G; Diabetes Outcome Progression Trial (ADOPT) Study Group. Rosiglitazone-associated fractures in type 2 diabetes: an Analysis from A Diabetes Outcome Progression Trial (ADOPT). Diabetes Care. 2008 May;31(5):845-51. doi: 10.2337/dc07-2270. Epub 2008 Jan 25. PMID 18223031
- [Background] Cohen A. Fecal blood loss and plasma salicylate study of salicylsalicylic acid and aspirin. J Clin Pharmacol. 1979 Apr;19(4):242-7. doi: 10.1002/j.1552-4604.1979.tb01658.x. PMID 312297
- [Background] Esser N, Paquot N, Scheen AJ. Anti-inflammatory agents to treat or prevent type 2 diabetes, metabolic syndrome and cardiovascular disease. Expert Opin Investig Drugs. 2015 Mar;24(3):283-307. doi: 10.1517/13543784.2015.974804. Epub 2014 Oct 25. PMID 25345753
- [Background] Ridker PM, Luscher TF. Anti-inflammatory therapies for cardiovascular disease. Eur Heart J. 2014 Jul 14;35(27):1782-91. doi: 10.1093/eurheartj/ehu203. Epub 2014 May 26. PMID 24864079
- [Background] Alderete TL, Sattler FR, Richey JM, Allayee H, Mittelman SD, Sheng X, Tucci J, Gyllenhammer LE, Grant EG, Goran MI. Salsalate treatment improves glycemia without altering adipose tissue in nondiabetic obese hispanics. Obesity (Silver Spring). 2015 Mar;23(3):543-51. doi: 10.1002/oby.20991. Epub 2015 Feb 3. PMID 25644856
- [Background] Pierce GL, Lesniewski LA, Lawson BR, Beske SD, Seals DR. Nuclear factor-kappaB activation contributes to vascular endothelial dysfunction via oxidative stress in overweight/obese middle-aged and older humans. Circulation. 2009 Mar 10;119(9):1284-92. doi: 10.1161/CIRCULATIONAHA.108.804294. Epub 2009 Feb 23. PMID 19237660
- [Background] Fleischman A, Shoelson SE, Bernier R, Goldfine AB. Salsalate improves glycemia and inflammatory parameters in obese young adults. Diabetes Care. 2008 Feb;31(2):289-94. doi: 10.2337/dc07-1338. Epub 2007 Oct 24. PMID 17959861
- [Background] Barzilay JI, Jablonski KA, Fonseca V, Shoelson SE, Goldfine AB, Strauch C, Monnier VM; TINSAL-T2D Research Consortium. The impact of salsalate treatment on serum levels of advanced glycation end products in type 2 diabetes. Diabetes Care. 2014 Apr;37(4):1083-91. doi: 10.2337/dc13-1527. Epub 2013 Nov 19. PMID 24255104
- [Background] Faghihimani E, Aminorroaya A, Rezvanian H, Adibi P, Ismail-Beigi F, Amini M. Salsalate improves glycemic control in patients with newly diagnosed type 2 diabetes. Acta Diabetol. 2013 Aug;50(4):537-43. doi: 10.1007/s00592-011-0329-2. Epub 2011 Sep 22. PMID 21938543
- [Background] Goldfine AB, Silver R, Aldhahi W, Cai D, Tatro E, Lee J, Shoelson SE. Use of salsalate to target inflammation in the treatment of insulin resistance and type 2 diabetes. Clin Transl Sci. 2008 May;1(1):36-43. doi: 10.1111/j.1752-8062.2008.00026.x. PMID 19337387
- [Background] Liang W, Verschuren L, Mulder P, van der Hoorn JW, Verheij J, van Dam AD, Boon MR, Princen HM, Havekes LM, Kleemann R, van den Hoek AM. Salsalate attenuates diet induced non-alcoholic steatohepatitis in mice by decreasing lipogenic and inflammatory processes. Br J Pharmacol. 2015 Nov;172(22):5293-305. doi: 10.1111/bph.13315. Epub 2015 Oct 22. PMID 26292849
- [Background] Goldfine AB, Fonseca V, Jablonski KA, Chen YD, Tipton L, Staten MA, Shoelson SE; Targeting Inflammation Using Salsalate in Type 2 Diabetes Study Team. Salicylate (salsalate) in patients with type 2 diabetes: a randomized trial. Ann Intern Med. 2013 Jul 2;159(1):1-12. doi: 10.7326/0003-4819-159-1-201307020-00003. PMID 23817699